CLINICAL TRIAL: NCT02902705
Title: Morphological and Functional Changes in White Adipose Tissue in Nondiabetic Chronic Kidney Disease Patients
Brief Title: Adipose Tissue & Uremia
Acronym: MODAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008.520
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease - Stage V
Keywords: White adipose tissue; chronic kidney disease; uremia; adipocytes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Kidney disease patients - stage V (Experimental): Male adults non-diabetic and non-dialyzed CKD stage 5 patients. All the CKD patient will be recruited at the Department of Nephrology of Edouard Herriot University Hospital (Lyon, France).
  Interventions: Other: Biopsy of abdominal subcutaneous white adipose tissue (2-3 g)
- Non Chronic Kidney Disease patients (Other): Non CKD male adults matched for age, gender and body mass index (BMI) with CKD patients. All the non - CKD patient will recruited from Department of recruited at the Department of Urology of Edouard Herriot University Hospital (Lyon, France).
  Interventions: Other: Biopsy of abdominal subcutaneous white adipose tissue (2-3 g)

INTERVENTIONS:
Other: Biopsy of abdominal subcutaneous white adipose tissue (2-3 g) — The biopsies of abdominal subcutaneous white adipose tissue (2-3 g) will be performed during elective surgery (i.e. peritoneal dialysis catheter) for CDK patients or during elective urologic surgery (e.g. radical prostatectomy) for Non-CDK patients. 50-100 mg will fixed in osmium tetroxide for cellularity measurement and 1g of fresh adipose tissue were used from adipocyte isolation. The remnant part of the biopsies will be snap frozen in liquid nitrogen and stored at -80°C until use (gene expression).

SUMMARY:
Many metabolic disturbances, such as protein-energy wasting, inulin resistance, and dyslipidemia are common features of chronic kidney disease (CKD). However, to date, the underlying mechanisms of these disturbances remain elusive. Many in vitro studies have demonstrated that white adipose cells exhibit dysfunctions in conditions that mimics uremic environment. In good agreement, several animal experiments have reported that chronic kidney disease was associated with lipoatrophy, adipose tissue dysfunction and ectopic lipid redistribution. The goal of this protocol is to collect and study structural and metabolic properties of white adipose tissue in CKD stage V patients to evidence adipose tissue dysfunction associated with CKD. The primary outcome measure will be the cellularity of the adipose tissue (i.e. size of the adipose cells) and the secondary measure to study the gene expression profile using microarray and metabolic properties of adipose tissue (i.e. lipogenesis). To this end, 15 male adult volunteers and 15 non-diabetic and non-dialyzed CKD stage V patients, matched for age, gender and body mass index (BMI) will be recruited at the Departments of Nephrology or Urology of Lyon University Hospital (Lyon, France). The biopsies of abdominal subcutaneous white adipose tissue (2-3 g) will be performed during elective urologic surgery (i.e. peritoneal dialysis catheter for CKD patients and radical prostatectomy for non CKD patients).

ELIGIBILITY:
Inclusion Criteria:

CKD (Chronic Kidney Disease) and non-CKD patients:

* At least 18 years of age
* Able and willing to provide informed consent
* Male gender
* Normal fasting glucose (less than 6 mmol/l )
* No evidence of significant concurrent illness
* BMI <30 kg/m2
* Non acidotic (bicarbonate >20 mmol/L)
* Normal coagulation profile

CKD patients:

• eGFR (estimated Glomerular Filtration Rate)< 25 mL/min/m2 before the beginning of renal suppletion therapy

Non-CKD patients:

• eGFR >50 mL/min/m2

Exclusion Criteria:

* A known diagnosis of diabetes mellitus
* enrolled in a other study that may confound results of this study.
* Have been treated with: corticosteroids or insulin or oral diabetic medications within 8 days prior to study entry
* Unwilling and/or not able to give written consent
* Patient with active systemic bacterial, viral or fungal infections

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Mean adipocyte size (in µm) in subcutaneous white adipose tissue removed during biopsy, measured with a Beckman Coulter | Day 1, the day of surgery (one day after inclusion)
  The biopsies of abdominal subcutaneous white adipose tissue (2-3 g) will be performed during elective surgery (i.e. peritoneal dialysis catheter for CKD patients and radical prostatectomy for non CKD patients). 50-100 mg will be fixed in osmium tetroxide for cellularity measurement i.e. measurement of adipose cell size. Adipose cell size will be determined by a Beckman Coulter Multisizer IV (Beckman Coulter) with a 400 µm aperture. The range of cell sizes that can effectively be measured using this aperture is 20-240 µm. The instrument will be set to count 1,000 particles, and the fixed-cell suspension will be diluted so that coincident counting remains <10%. Cell-size distributions will be drawn from measurement of at least 12,000 cell diameters for each patient. The mean fat cell volume will then be compared using Student t test or Mann & Whitney U tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie, dialyse, hypertension artérielle - Pavillon P - Hôpital Edouard Herriot -, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luce M, Barba C, Yi D, Mey A, Roussel D, Bres E, Benoit B, Pastural M, Granjon S, Szelag JC, Laville M, Arkouche W, Bouchara A, Nyam E, Fouque D, Soulage CO, Koppe L. Accumulation of natriuretic peptides is associated with protein energy wasting and activation of browning in white adipose tissue in chronic kidney disease. Kidney Int. 2020 Sep;98(3):663-672. doi: 10.1016/j.kint.2020.03.027. Epub 2020 Apr 23. PMID 32739210